CLINICAL TRIAL: NCT04620460
Title: Efficacy and Mechanisms of Low-intensity Focused Ultrasound on Negative Symptoms in Patients With Schizophrenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Principal Investigator, Dengtang LIU, Chief Psychiatrist and Professor, Shanghai Mental Health Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-TX-006
Record Dates: First submitted 2020-10-15; First posted 2020-11-09 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Negative Symptoms of Schizophrenia
Keywords: Low-intensity Focused Ultrasound; Negative Symptoms of Schizophrenia Patients

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LIFUS-left DLPFC (Active Comparator): 20 patients will be treated with active LIFUS for 3 weeks on the left DLPFC.
  Interventions: Device: Low-intensity Focused Ultrasound(LIFUS)
- LIFUS-SHAM (Sham Comparator): 20 patients will be treated with sham LIFUS for 3 weeks on the left DLPFC.
  Interventions: Device: Low-intensity Focused Ultrasound(LIFUS)

INTERVENTIONS:
Device: Low-intensity Focused Ultrasound(LIFUS) — Patients with schizophrenia will be treated with active LIFUS or sham stimulation for 3 weeks on the left DLPFC.

SUMMARY:
Based on our research background, we hypothesize that LIFUS has neuromodulation effects on brain cortex and the active LIFUS on left-DLPFC would improve negative symptoms in schizophrenia patients. It would firstly verify the safety of LIFUS on human as well. The multimodal MRI will be contributed to investigate the possible mechanism of negative symptoms.

DETAILED DESCRIPTION:
Firstly, we plan to explore the short-term effects of LIFUS on cortical excitability by detecting the MEP amplitude. 40 patients and relatively well matched healthy-control would be enrolled. After MEP detection and baseline evaluations, the two groups will be treated with one-single intervention on the primary motor cortex. The cognitive function and MEP amplitude will be assessed respectively at the moment, after 15 minutes and 30 minutes. Then, it is a randomized double-blind sham-controlled LIFUS intervention trial in schizophrenia patients. After screening and baseline evaluations, the 40 patients with schizophrenia will be treated with active LIFUS or sham stimulation for 3 weeks on the left DLPFC. The multimodal MRI will be acquired. Clinical symptoms and cognitive function will be assessed respectively at baseline, at the end of fifth treatments and after the end of the treatment.

ELIGIBILITY:
* Inclusion Criteria (patients):

  1. Meet the DSM-5 diagnostic criteria for schizophrenia or schizoaffective disorder;
  2. Age18-50, right-handed, Han nationality;
  3. the score of at least 1 item from N1 to N7 is ≥4 (moderate or above);
  4. Be in a stable condition, received second-generation antipsychotics for at least 4 weeks or more;
  5. Written informed consent;
* Exclusion Criteria (patients):

  1. Current or past neurological illness, severe physical diseases, substance abuse or alcohol dependence, mental retardation, pregnant or lactation;
  2. Uncooperative or risky patients with high excitement, stupor, disorder of words and deeds, negative suicide, etc.;
  3. A history of MECT or other physical therapy within 6 months;
  4. A history of epilepsy, or epileptic waves on the baseline EEG;
  5. Ruled out share antiepileptic drugs, carbamazepine, valproic acid salt) or larger doses of benzodiazepines drugs (> 10 mg/day, diazepam clonazepam 2 mg/day, 1 mg/day, alprazolam lorazepam 2 mg/day, midazolam 10 mg/day, 20 mg/day, Mr Shah diazepam triazolam 0.5 mg/day), avoid the use of chlorine drug, (in principle, to avoid the use of antiepileptic drugs and clonazepam;Other antipsychotic drugs, if necessary, remain unchanged during the course of treatment;
  6. Contraindications to LIFUS and MRI are present.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-08-05 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Clinical Symptoms-PANSS | baseline and 15 days
  Change from baseline in Positive and Negative Syndrome Scale(PANSS)
Clinical Symptoms-SANS | baseline and 15 days
  Change from baseline in the Scale for the Assessment of Negative Symptoms(SANS)

SECONDARY OUTCOMES:
Cognitive Function | baseline, after the fifth treatment and 15 days
  Change from baseline in the Brief Cognition Test (C-BCT)
Change of brain neuroimaging | baseline, fifth treatment and 15th treatment
  Brain structure, Resting-state fMRI data, Arterial Spin Labeling(ASL), 1H-MRS in DLPFC are acquired.
Cortex Excitability | baseline，the moment after the intervention, after 15 minutes and 30 minutes
  MEP amplitude

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhai Z, Ren L, Song Z, Xiang Q, Zhuo K, Zhang S, Li X, Zhang Y, Jiao X, Tong S, Sun J, Liu D. The efficacy of low-intensity transcranial ultrasound stimulation on negative symptoms in schizophrenia: A double-blind, randomized sham-controlled study. Brain Stimul. 2023 May-Jun;16(3):790-792. doi: 10.1016/j.brs.2023.04.021. Epub 2023 Apr 29. No abstract available. PMID 37121354